CLINICAL TRIAL: NCT02133183
Title: Pilot Study of MLN0128 (TAK-228) in Preoperative Recurrent Glioblastoma (GBM) Patients
Brief Title: Sapanisertib Before and After Surgery in Treating Patients With Recurrent Glioblastoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Other - Lapse in funding
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-00907; NCI-2014-00907 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ABTC-1301; 1301; ABTC-1301 (Other: Adult Brain Tumor Consortium); ABTC-1301 (Other: CTEP); U01CA137443 (NIH); UM1CA137443 (NIH)
Record Dates: First submitted 2014-05-06; First posted 2014-05-07 (Estimated); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Glioblastoma; Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — sapanisertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (sapanisertib before and after surgery) (Experimental): Patients receive sapanisertib PO according to the results from Part I. Patients also undergo surgery on day 0. Within 45 days after surgery, patients receive sapanisertib PO according to the results from Part I. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Sapanisertib; Procedure: Therapeutic Conventional Surgery
- Arm II (sapanisertib after surgery) (Experimental): Patients undergo surgery on day 0. Within 45 days after surgery, patients receive sapanisertib PO according to the results from Part I. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Sapanisertib; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Sapanisertib — Given PO
  Other Names: INK-128; INK128; MLN-0128; MLN0128; TAK-228
Procedure: Therapeutic Conventional Surgery — Undergo surgery

SUMMARY:
This partially randomized pilot phase I trial studies how much sapanisertib reaches the brain tumor and how well it works when given before and after surgery in treating patients with glioblastoma that has grown or come back and requires surgery. Sapanisertib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the penetration of sapanisertib (MLN0128 [TAK-228]) across the blood brain barrier and achieve a concentration of 70 nM in tissue resected from a contrast enhancing region of the tumor in 60% of recurrent glioblastoma (GBM) patients. (Part I) II. To determine the ability of MLN0128 (TAK-228) to inhibit TOR complex (TORC)1/2 in the enhancing components of the tumor as determined by modulation of RPS6 phosphorylated Ser-235 (pS235) in reverse phase protein array (RPPA) assays. (Part II)

SECONDARY OBJECTIVES:

I. To evaluate the penetration of MLN0128 (TAK-228) across the blood brain barrier by determining its concentration in tissue resected from a non-contrast enhancing region of the tumor. (Part I) II. To assess the plasma pharmacokinetics of MLN0128 (TAK-228) in patients with recurrent GBM. (Part I) III. To determine the ability of MLN0128 (TAK-228) to inhibit TORC1/2 in the non-enhancing components of the tumor as determined by modulation of RPS6 pS235 in RPPA assays. (Part II) IV. To assess the ability of MLN0128 (TAK-228) to inhibit TORC1/2 by evaluating pharmacodynamics (PD) markers by immunohistochemistry such as pS235, pS236, phosphorylated 4E-binding protein (p4EBP), phosphorylated-mechanistic target of rapamycin (serine/threonine kinase) (pmTOR), and AKTpSer473. (Phase II) V. To evaluate the safety profile of MLN0128 (TAK-228) in pre-operative patients with recurrent GBM.

VI. To estimate response rate, progression-free survival, and overall survival.

TERTIARY OBJECTIVES:

I. To perform mass spectrometry imaging (MSI) to qualitatively assess the ability of MLN0128 (TAK-228) to penetrate the blood brain barrier and enter tumor tissue in enhancing and non-enhancing regions of the tumor. (Part I) II. To determine ex-vivo sensitivity of tumor neurosphere cultures (patient derived cell lines [PDCL]) established from surgical specimens to MLN0128 (TAK-228). (Part II) III. To explore the potential association of tumor genotype with progression-free survival among patients treated with MLN0128 (TAK-228). (Part II) IV. To determine the ability of MLN0128 (TAK-228) to inhibit TORC1/2 as determined by modulation of additional TORC1/2 markers in RPPA assays. (Part II)

OUTLINE:

PART I:

COHORT A: Patients receive sapanisertib orally (PO) once daily (QD) for 7-9 days (including 2-4 hours before surgery). On day 0, patients undergo surgery. Within 45 days after surgery, patients receive sapanisertib PO QD. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. If patients do not demonstrate adequate sapanisertib tumor tissue concentrations, patients are enrolled in Cohort B.

COHORT B: Patients receive sapanisertib PO 2-4 hours before surgery on day 0. Within 45 days after surgery, patients receive sapanisertib PO once weekly. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

PART II: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive sapanisertib PO according to the results from Part I. Patients also undergo surgery on day 0. Within 30 days after surgery, patients receive sapanisertib PO according to the results from Part I. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients undergo surgery on day 0. Within 30 days after surgery, patients receive sapanisertib PO according to the results from Part I. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, every 2 months for 2 years, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically proven glioblastoma or gliosarcoma which is progressive or recurrent following radiation therapy +/- chemotherapy
* Patients must have measurable, supratentorial contrast-enhancing progressive or recurrent glioblastoma or gliosarcoma by magnetic resonance imaging (MRI) imaging within 21 days of starting treatment; patient must be able to tolerate MRIs
* Patients may have had treatment for no more than 2 prior relapses
* Patients must have recovered from severe toxicity of prior therapy; the following intervals from previous treatments are required to be eligible:

  * 12 weeks from the completion of radiation
  * 6 weeks from a nitrosourea chemotherapy or mitomycin C
  * 3 weeks from a non-nitrosourea chemotherapy
  * 4 weeks from any investigational (not Food and Drug Administration [FDA]-approved) agents
  * 2 weeks from administration of a non-cytotoxic, FDA-approved agent except bevacizumab/vascular endothelial growth factor receptor (VEGFR) inhibitors (e.g., erlotinib, hydroxychloroquine, etc.)
  * 6 weeks from bevacizumab/VEGFR inhibitors
* Patients must be undergoing surgery that is clinically indicated as determined by their care providers
* Patients must be eligible for surgical resection according to the following criteria:

  * Part 1 Patients: Expectation that the surgeon is able to resect at least 350 mg of tumor from enhancing tumor and at least 350 mg from non-enhancing tumor with low risk of inducing neurological injury
  * Part 2 Patients: Expectation that the surgeon is able to resect at least 1000 mg from enhancing tumor and at least 350 mg from non-enhancing tumor with low risk of inducing neurological injury
* Patients must have a Karnofsky performance status >= 60% (i.e. the patient must be able to care for himself/herself with occasional help from others)
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Fasting serum glucose =< 130 MG/DL
* HbA1c =< 7.0%
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 × institutional upper limit of normal
* Creatinine =< institutional upper limit of normal OR
* Creatinine clearance >= 50 ml/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Activated partial thromboplastin time (APTT)/partial thromboplastin time (PTT) =< 1.5 x institutional upper limit of normal
* Patients must be able to provide written informed consent
* Women of childbearing potential must have a negative serum pregnancy test prior to study entry; women of childbearing potential and men must agree to practice 1 highly effective method of contraception and 1 additional effective (barrier) method, at the same time, prior to study entry, for the duration of study participation, and through 90 days (or longer, as mandated by local labeling [e.g. USPI, SmPC, etc.]) after the last dose of study drug; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use highly effective barrier contraception prior to the study, for the duration of study participation, and through 120 days after the last dose of study drug
* Patients must have no concurrent malignancy except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix, breast, or bladder; patients with prior malignancies must be disease-free for >= five years
* Patients must be able to swallow whole capsules
* Patients enrolled in Part 2 must have at least 20 (preferably 40) slides of archival tumor tissue from a prior surgery demonstrating GBM; patients enrolled in Part 1 will not be required to have archival tissue
* Patients with controlled diabetes are allowed on study; controlled diabetes is defined as < 130 ml/dL for the sake of this study

Exclusion Criteria:

* Patients receiving any other investigational agents are ineligible
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to MLN0128 (TAK-228) are ineligible
* Patients may not have had prior treatment with mTOR, peptidase inhibitor 3, skin-derived (PI3) kinase or Akt inhibitors
* Patients on enzyme-inducing anti-epileptic drugs (EIAED) are not eligible for treatment on this protocol; patients may be on non-enzyme inducing anti-epileptic drugs or not be taking any anti-epileptic drugs; patients previously treated with EIAED may be enrolled if they have been off the EIAED for 10 days or more prior to the first dose of MLN0128 (TAK-228)
* Patients must not have evidence of significant hematologic, renal, or hepatic dysfunction
* Patients must not have evidence of significant intracranial hemorrhage
* Patients with a history of any of the following within the last 6 months prior to study entry are ineligible:

  * Ischemic myocardial event, including angina requiring therapy and artery revascularization procedures
  * Ischemic cerebrovascular event, including transient ischemic attack (TIA) and artery revascularization procedures
  * Requirement for inotropic support (excluding digoxin) or serious (uncontrolled) cardiac arrhythmia (including atrial flutter/fibrillation, ventricular fibrillation or ventricular tachycardia)
  * Placement of a pacemaker for control of rhythm
  * New York Heart Association (NYHA) class III or IV heart failure
  * Pulmonary embolism
* Patients with known significant active cardiovascular or pulmonary disease at the time of study entry are ineligible
* Patients with baseline prolongation of the rate-corrected QT interval (QTc) (e.g., repeated demonstration of QTc interval > 480 milliseconds, or history of congenital long QT syndrome, or torsades de pointes) are ineligible
* Patients with known diabetes mellitus which is poorly controlled (defined as hemoglobin A1c [HbA1c] > 7%) are ineligible; subjects with a history of transient glucose intolerance due to corticosteroid administration are allowed in this study if all other inclusion/exclusion have been met
* Patients who have initiated treatment with bisphosphonates less than 30 days prior to the first administration of MLN0128 (TAK-228) are ineligible; concurrent bisphosphonate use is only allowed if the bisphosphonate was initiated at least 30 days prior to the first administration of MLN0128 (TAK-228)
* For weekly MLN0128 (TAK-228) dose cohorts, patients taking proton pump inhibitors (PPIs) are ineligible unless these patients are able to switch to a histamine (H2) blocker and/or antacid
* Patients with known manifestations of malabsorption due to prior gastrointestinal (GI) surgery, GI disease, or for an unknown reason that may alter the absorption of MLN0128 (TAK-228) are ineligible
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements, are ineligible
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with this agent
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Subjects taking strong CYP3A4 and CYP2C19 inhibitors and/or inducers should be considered with caution; alternative treatments that are less likely to affect MLN0128 (TAK-228) metabolism, if available, should be considered; if a subject requires treatment with 1 or more of the strong CYP3A4 and CYP2C19 inhibitors and/or inducers, the study doctor should be consulted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-07-02 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who achieve a drug concentration >= 70 nM in contrast enhancing tumor tissue | Up to 2 years
  The proportion of patients who achieve a drug concentration >= 70 nM in contrast enhancing tumor tissue will be calculated and the 90% confidence interval will be estimated using binomial distribution.
Difference in ratio of the S6 phosphorylation over the total between the two groups | Up to 2 years
  Two sample t-test will be used for the hypothesis testing of a difference in ratio of the S6 phosphorylation over the total between the two groups.
Difference of the pS6 concentration between the two groups | Up to 2 years
  Two sample t-test will be used for the hypothesis testing of a difference in ratio of the S6 phosphorylation over the total between the two groups. A "heat map" or "heat map visualization" may also be used to present and examine possible difference in clustering signaling pathway activation between the groups.

SECONDARY OUTCOMES:
Sapanisertib concentration in non-enhancing tumor | Up to 2 years
  Will be summarized using descriptive statistics or two-group comparison between groups. The Spearman correlation coefficient might be used to assess potential correlations between pathway modulation scores and tumor growth measured by KI67 (proliferation) and cleaved caspase 3 (apoptosis/cell death).
Sapanisertib concentration in blood | Up to 2 years
  Will be summarized using descriptive statistics or two-group comparison between Groups A and B. The Spearman correlation coefficient might be used to assess potential correlations between pathway modulation scores and tumor growth measured by KI67 (proliferation) and cleaved caspase 3 (apoptosis/cell death).
Inhibition TORC1/2 in the non-enhancing components of the tumor as determined by modulation of RPS6 pS235 in reverse phase protein array (RPPA) assays | Up to 2 years
  Will be summarized using descriptive statistics or two-group comparison between Groups A and B. The Spearman correlation coefficient might be used to assess potential correlations between pathway modulation scores and tumor growth measured by KI67 (proliferation) and cleaved caspase 3 (apoptosis/cell death).
Pharmacodynamic marker such as pS6 (by immunohistochemistry), p4EBP, pmTOR, and AKTpSer473 compared to the control | Up to 2 years
  Will be summarized using descriptive statistics or two-group comparison between Groups A and B. The Spearman correlation coefficient might be used to assess potential correlations between pathway modulation scores and tumor growth measured by KI67 (proliferation) and cleaved caspase 3 (apoptosis/cell death).
Incidence of toxicity graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 | Up to 30 days
  All treatment or surgically related adverse events will be reported descriptively. A proportion of toxicity grade >= 3 will be estimated using binomial distribution.
Tumor response | Up to 2 years
  The proportion of patients who had tumor response (partial response + complete response) during the course of treatment will be estimated using the exact binomial distribution.
Progression-free survival (PFS) | Time from date of post-surgical treatment start to the date progressive disease was defined, assessed up to 2 years
  PFS along with 95% confidence interval will be estimated using Kaplan-Meier method.
Overall survival (death) | Time from the date of post-surgical treatment start to the date death occurred, assessed up to 2 years
  Overall survival along with 95% confidence interval will be estimated using Kaplan-Meier method.

OTHER OUTCOMES:
MSI from treated versus (vs) untreated enhancing and non- enhancing tumor | Up to 2 years
  MSI from treated vs untreated enhancing and non- enhancing tumor will be compared using visualization and presented by graph and descriptive statistics.
Ex-vivo sensitivity of tumor sphere cultures established from surgical specimens to sapanisertib, defined by a minimum of 20% reduction in cell proliferation as measured by cell titer glow in the sapanisertib group compared to the untreated group | Up to 2 years
  Fisher's exact test will be used for testing a difference in the proportion between the two groups.
Tumor genotype | Up to 2 years
  Cox regression model or logistic regression model will be used to explore associations between PD outcome or tumor genotype and overall survival or progression-free survival. All estimated associations will be reported along with 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Eudocia Q Lee, Principal Investigator — National Cancer Institute (NCI)
Locations (10):
- United States (10):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Arnold A, Rodriguez F, Eberhart CG, Raabe EH. Response to letter to the editor: "All models are wrong; some models are useful". Neuro Oncol. 2020 Sep 29;22(9):1406-1407. doi: 10.1093/neuonc/noaa137. No abstract available. PMID 32597469